CLINICAL TRIAL: NCT05662657
Title: Prevalence of Post Traumatic Stress Disorder Related to Diabetes Diagnosis or Severe Hypoglycaemia in Adult With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Sponsor
Other Study IDs: DIASPOT
Record Dates: First submitted 2022-12-02; First posted 2022-12-22 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: PCL-S Questionnaire — PCL-S and HADS questionnaires
  Other Names: Diagnostic Test: HADS Questionnaire

SUMMARY:
In France, the adult population living with diabetes in 2016 is estimated at more than 3.3 million patients treated. Type 1 diabetes (T1DM) represents 5.6% of diabetic patients (approximately 185,000 patients).

Numerous studies show that patients fear hypoglycemia, with an impact on their quality of life, sleep disorders and depressive symptoms. In addition, there is a metabolic impact with a problem of therapeutic compliance and an alteration of glycemic control.

This study examine the relation between Post Traumatic Stress disorder (PTSD) and diabetes diagnosis or severe hypoglycaemia in adults with Type 1 Diabetes.

The aim of this study is to evaluate the prevalence of PTSD in this population.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* With type 1 diabetes,
* Willing and able to complete all the questionnaires in French,
* Who have given oral consent,
* being affiliated to a social security scheme or being a beneficiary of such a scheme.

Exclusion Criteria:

* Non-diabetic type 1,
* With an unstable psychiatric pathology,
* Pregnant or breastfeeding women,
* Subject to a measure for the protection of justice,
* Having opposed the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: population of insulin-treated type 1 diabetic patients
Sampling Method: Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
To evaluate the prevalence of post-traumatic stress disorder (PTSD) in adult with Type 1 Diabetes | baseline
  Score (>44) measured on the Posttraumatic Stress Disorder Checklist Scale (PCL-S) for severe hypoglycemia

SECONDARY OUTCOMES:
To evaluate the prevalence of post-traumatic stress disorder (PTSD). This PTSD is related to diabetes diagnosis and its initial management. | baseline
  Score (>44) measured on the Posttraumatic Stress Disorder Checklist Scale (PCL-S).
  The patient will complete the questionnaire once to evaluate PTSD related to both diabete diagnosis and its initial management.
To evaluate the prevalence of post-traumatic stress disorder (PTSD) related to severe hypoglycemia. | baseline
  Score (>44) measured on the Posttraumatic Stress Disorder Checklist Scale (PCL-S) for severe hypoglycemia
To evaluate the prevalence of post-traumatic stress disorder (PTSD). This PTSD is related to at least one of the following reasons : - severe hypoglycemia - diabetes diagnosis and its initial management. | baseline
  Score (>44) measured on the Posttraumatic Stress Disorder Checklist Scale (PCL-S).
  The patient will complete the questionnaire once to evaluate PTSD related to severe hypoglycemia and/or diabetes diagnosis and its initial management
To evaluate the prevalence of anxiety-depressive disorder in adults with type 1 diabetes | baseline
  Score (from 0 to 42 ) measured on the Hospital Anxiety and Depression Scale (HADS)
  Total scores can be categorized into five levels:
  * HADS score of 7 or less = no symptoms,
  * HADS score of 8 to 10 = doubtful symptomatology,
  * HADS score of 11 or more = definite symptomatology.
To demonstrate the presence of anxiety-depressive disorder related to PTSD | baseline
  Rate of patients with anxiety depressive disorder associated with PTSD
To evaluate whether there is a correlation between PTSD and the patient participation to a therapeutic education program | baseline
  Percentage of patients with PTSD (PCL-S > 44) between groups of patients participating or not in a therapeutic education program (Functional Insulin Therapy or multidisciplinary education in day hospital or hospitalization)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopital Saint Joseph, Marseille
  - Centre Hospitalier de Martigues, Martigues

IPD SHARING:
Plan to Share IPD: No
The participants of this study did not give written consent for their data to be shared publicly, so due to the sensitive nature of the research supporting data is not available